CLINICAL TRIAL: NCT05860153
Title: Intermittent Levetricetam in Treatment of Febrile Convulsions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kariman Hussein Tawfik, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Febrile convulsions treatment
Record Dates: First submitted 2023-04-18; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Febrile Convulsion
MeSH Terms: conditions — Seizures, Febrile | interventions — Levetiracetam; Diazepam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): • Group (A) will receive oral levetiracetam at a dose of 15-20 mg/kg/day twice daily at the onset of fever (temperature >37.5 c) for 48h after subsiding of fever.
  Interventions: Drug: Levetiracetam
- Group (B) (Experimental): • Group (B) will receive diazepam at a dose of 0.3 mg/kg/dose was given every eight hours for 48h after subsiding of fever Children were followed up for 12 months to find out seizure frequency associated with febrile events and febrile seizure recurrence rate during 12 months follow-up
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Levetiracetam — Group with oral levetiracetam at a dose of 15-20 mg/kg/day
  Other Names: Tiratam
  Arms: Group (A)
Drug: Diazepam — Group with diazepam at a dose of 0.3 mg/kg/dose
  Other Names: Valinil
  Arms: Group (B)

SUMMARY:
The American Academy of Pediatrics (AAP) in 2011 published a clinical practice guideline defining a febrile seizure as "a seizure accompanied by fever (temperature ≥ 100.4°F or 38°C by any method), without central nervous system infection, that occurs in infants and children 6 through 60 months of age." Febrile seizures are further classified as simple (generalized in onset, last less than 15 minutes, and do not occur more than once in 24 hours.) or complex (FS duration longer than 15 min, repeated convulsions within the same day, and focal seizure activity or focal findings during the postictal period.).

DETAILED DESCRIPTION:
The American Academy of Pediatrics (AAP) in 2011 published a clinical practice guideline defining a febrile seizure as "a seizure accompanied by fever (temperature ≥ 100.4°F or 38°C by any method), without central nervous system infection, that occurs in infants and children 6 through 60 months of age." Febrile seizures are further classified as simple (generalized in onset, last less than 15 minutes, and do not occur more than once in 24 hours.) or complex (FS duration longer than 15 min, repeated convulsions within the same day, and focal seizure activity or focal findings during the postictal period.).

Epidemiology Approximately 8% of people will experience at least one seizure episode during their lifetime. Up to 30% of such episodes are febrile seizures (FS), which are the most commonly occurring seizures in 2 to 5% of all children. Nevertheless, although FS is a benign condition in most cases and the prognosis is good generally and recurrences do not impair the prognosis in children who were neurologically normal before their first febrile seizure, FS episodes constitute a traumatic experience, it is a very frightening event for the parents/caregivers witnessing a tonic-clonic seizure, especially for the patients with frequent FS, they suffer extreme anxiety for recurrences of seizures or development of epilepsy; FS is also likely one of the most frequent causes of admittance to pediatric emergency ward worldwide. In any case, febrile seizures should be taken under serious consideration.

During seventies ten eligible clinical trials were included. Prophylaxis with either phenobarbital or diazepam reduces recurrences of febrile seizures.

After oral administration >90% of diazepam is absorbed and the average time to achieve peak plasma concentrations is 1 - 1.5 hours with a range of 0.25 to 2.5 hours. The mean half-life of diazepam has been reported to be 18 hours. Intermittent diazepam in oral or anal form is effective In preventing the recurrence of febrile seizures as diazepam however, the side effects associated with intermittent diazepam in the prevention of febrile seizures outweight it's potential benefits including sedation, behavioral changes, gastrointestinal and hematologic toxicity, hypersensitivity reactions, and rare fatal hepatotoxicity with VPA in young children. And also the intermittent administration of benzodiazepines (e.g., diazepam and midazolam) at the onset of fever is effective, but the effectiveness of this treatment is limited because sedative effects can mask the signs and symptoms of any evolving central nervous system infections.

After oral ingestion, levetiracetam is rapidly absorbed, with peak concentration occurring after 1.3 hours, and its bioavailability is ≥95%. LEV was reported to induce psychotropic side effects in up to 30% of patients. These adverse effects include beneficial effects such as enhancement of drive and cognition on the one hand and behavioral disturbances such as irritability, aggression, agitation, anger, anxiety, apathy, and hostility on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* Included children 6 months to 36 months with febrile seizures after exclusion of CNS infections .

Exclusion Criteria:

* Non-febrile seizures
* Head trauma
* CNS infections
* Known metabolic diseases
* Known genetic disorders
* Developmental delay

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of therapeutic effect of oral levetiracetam on febrile convulsions | Baseline
  The rate of therapeutic effect of oral levetiracetam in reducing the recurrence of febrile seizures in children aged 6-36months.
The rate of therapeutic effect of intermittent diazepam on febrile convulsions | Baseline
  The rate of therapeutic effect of intermittent diazepam in reducing the recurrence of febrile seizures in children aged 6-36months.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Elsayah, Prof, Principal Investigator — Assiut University; Khalaf Abd El-Aal, Assist prof, Principal Investigator — Assiut University